CLINICAL TRIAL: NCT06593327
Title: Evaluation of a Pragmatic NT-ProBNP-based Heart Failure Screening Strategy Among Patients with Type 2 Diabetes: STRONG-DM Study (Screening and Treatment Using Risk-based ApprOach with NT-ProBNP Guidance in Diabetes Mellitus
Brief Title: NT-ProBNP-based Heart Failure Screening and Prevention Trial in Patients with Type 2 Diabetes: STRONG-DM Study
Acronym: STRONG-DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Principal Investigator, Ambarish Pandey, Associate Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU-2024-0458
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes; Diabetic Cardiomyopathy; Heart Failure; Cardiometabolic Diseases
Keywords: Pragmatic Clinical Trial; Heart Failure; Cardiovascular Prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Cardiomyopathies; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Risk Assessment and Intensive Prevention Strategy (Experimental): Primary care providers (PCP) randomized to the Risk Assessment and Intensive Prevention Strategy Arm will receive notification if any patients with diabetes under their care have high heart failure risk based on clinical or biomarker scores. Providers will receive recommendations, option for e-consultation, and referral to cardiometabolic risk management program.
  Interventions: Behavioral: Intensive Prevention Strategy
- Usual Care (No Intervention): Primary care providers randomized to the Usual care arm will not receive any notifications about patients with diabetes and their HF risk assessment.

INTERVENTIONS:
Behavioral: Intensive Prevention Strategy — Providers randomized to the intensive prevention strategy will receive notification about patients with diabetes who have high heart failure risk and recommendations for medical management, e-consultation, or referral to a cardiometabolic risk management program.
  Arms: Risk Assessment and Intensive Prevention Strategy

SUMMARY:
A pragmatic, randomized clinical trial to evaluate the effect of a heart failure (HF) risk assessment and prevention strategy incorporating HF clinical risk scores (WATCH-DM) with cardiac biomarker (NT-proBNP) paired with a clinical decision support tool to implement an intensive prevention strategy among patients with high risk focused on implementation of evidence-based HF preventive therapies.

DETAILED DESCRIPTION:
Primary care providers will be randomized to receive notifications via the electronic health record if any patients with diabetes have high heart failure risk based on a combination of clinical risk scores(WATCH-DM), and biomarkers (NT-proBNP). Providers will be provided recommendation to initiate evidence based therapies (SGLT2 inhibitors, GLP1 agonists, non-steroidal MRA) , obtain expert e-consultation, or refer the patient to a cardiometabolic risk management program.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care Provider that sees diabetes patients in clinic

Exclusion Criteria:

* Provider does not see patients with Diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-12-10 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Incident Heart Failure or All-cause death | 2-year follow-up
  Incident Heart Failure (based on electronic health record International Classification of Diseases codes) or all-cause death. This will be assessed via retrospective chart review.

SECONDARY OUTCOMES:
Prescription Rates of SGLT2i | 6-months from electronic health record alert.
  Counts of SGLT2 inhibitor prescriptions filled
Prescription Rate of Finerenone | 6-months from electronic health record alert.
  Counts of Finerenone prescriptions
Prescription Rate of GLP1 | 6-months from electronic health record alert.
  Counts of GLP1 prescription

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No